CLINICAL TRIAL: NCT04722887
Title: A Multi-Center, Single-Dose and Repeat-Dose Over Eight Weeks, Sequential Cohort Study to Evaluate Safety and Tolerability as Well as Pharmacokinetics of Two Different Doses of Alpha1-Proteinase Inhibitor Subcutaneous (Human) 15% Administered Subcutaneously in Subjects With Alpha1-Antitrypsin Deficiency
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of Two Different Doses of Alpha1-Proteinase Inhibitor Subcutaneous (Human) 15% in Participants With Alpha1-Antitrypsin Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC2008
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Alpha1-Antitrypsin Deficiency
Keywords: Pulmonary Emphysema; Alpha-1 Antitrypsin Deficiency; AATD; Alpha-1 PI Deficiency; Alpha-1 Proteinase Inhibitor; Emphysema; Pathologic Processes; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Lung Diseases; Respiratory Tract Diseases; Liver Diseases; Digestive System Diseases; Genetic Diseases, Inborn; Subcutaneous Emphysema; Alpha1-Antitrypsin; Trypsin Inhibitors; Serine Proteinase Inhibitors; Protease Inhibitors; Enzyme Inhibition; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Emphysema; Emphysema; Pathologic Processes; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Lung Diseases; Respiratory Tract Diseases; Liver Diseases; Digestive System Diseases; Genetic Diseases, Inborn; Subcutaneous Emphysema | interventions — 15-keto-17-phenyl-18,19,20-trinorprostaglandin F2 alpha-1-isopropyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Treatment Period 1 (Alpha-1 15%, 72 mg/kg) (Experimental): Participants will receive Alpha-1 15% 72 mg/kg, single weekly subcutaneous (SC) infusion in treatment-period 1 (Single-Dose) at Week 1.
  Interventions: Biological: Alpha-1 15%
- Cohort 1: Single-Dose Data Evaluation Period (Liquid Alpha 1-Proteinase Inhibitor 60 mg/kg) (Experimental): Following treatment period 1, participants in Cohort 1 will enter 21 days of washout/serial pharmacokinetic (PK) phase and then the single-dose data evaluation period. During the single-dose data evaluation phase, Liquid Alpha1- Proteinase Inhibitor (PI) 60 mg/kg, weekly intravenous (IV) Infusions will be administered from intravenous-dose Week 1 (single-dose Week 5) for up to Week 78, with the last IV dose given 1 week prior to the first repeat Alpha-1 15% SC dose.
  Interventions: Biological: Liquid Alpha1-Proteinase Inhibitor (Human)
- Cohort 1: Treatment Period 2 (Alpha-1 15%, 72 mg/kg) (Experimental): Following treatment period 1 and single-dose data evaluation period, participants in Cohort 1 will enter treatment period 2 (Repeat-Dose) and will receive Alpha-1 15% 72 mg/kg, for 8 weekly SC infusions.
  Interventions: Biological: Alpha-1 15%
- Cohort 2: Treatment Period 1 (Alpha-1 15%, 180 mg/kg) (Experimental): Participants will receive Alpha-1 15% 180 mg/kg, single weekly SC infusion in treatment-period 1 (Single-Dose) at Week 1.
  Interventions: Biological: Alpha-1 15%
- Cohort 2: Single-Dose Data Evaluation Period (Liquid Alpha1-Proteinase Inhibitor 120 mg/kg) (Experimental): Following treatment period 1, participants in Cohort 2 will enter 21 days of washout/serial pharmacokinetic (PK) phase and then the single-dose data evaluation phase. During the single-dose data evaluation phase, Liquid Alpha1-PI 120 mg/kg, weekly IV Infusions will be administered from intravenous-dose Week 1 (single-dose Week 5) for up to Week 78, with the last IV dose given 1 week prior to the first repeat Alpha-1 15% SC dose.
  Interventions: Biological: Liquid Alpha1-Proteinase Inhibitor (Human)
- Cohort 2: Treatment Period 2 (Alpha-1 15%, 180 mg/kg) (Experimental): Following treatment period 1 and single-dose data evaluation phase, participants in Cohort 2 will enter treatment period 2 (Repeat-Dose) and will receive Alpha-1 15% 180 mg/kg, for 8 weekly SC infusions.
  Interventions: Biological: Alpha-1 15%

INTERVENTIONS:
Biological: Alpha-1 15% — Alpha1-Proteinase Inhibitor (Human), 15%, Subcutaneous infusion
  Arms: Cohort 1: Treatment Period 1 (Alpha-1 15%, 72 mg/kg); Cohort 1: Treatment Period 2 (Alpha-1 15%, 72 mg/kg); Cohort 2: Treatment Period 1 (Alpha-1 15%, 180 mg/kg); Cohort 2: Treatment Period 2 (Alpha-1 15%, 180 mg/kg)
Biological: Liquid Alpha1-Proteinase Inhibitor (Human) — Intravenous infusion
  Other Names: Prolastin®-C Liquid
  Arms: Cohort 1: Single-Dose Data Evaluation Period (Liquid Alpha 1-Proteinase Inhibitor 60 mg/kg); Cohort 2: Single-Dose Data Evaluation Period (Liquid Alpha1-Proteinase Inhibitor 120 mg/kg)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of 72 milligrams per kilogram (mg/kg) and 180 mg/kg Alpha-1 15%, administered as a single-dose subcutaneous (SC) infusion and subsequently as weekly SC infusions over 8 weeks in participants with Alpha1-Antitrypsin Deficiency (AATD).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of congenital Alpha1-antitrypsin deficiency (AATD) with an allelic combination of ZZ, SZ, Z(null), (null)(null), S(null), or "at-risk" alleles (subjects with "at-risk" alleles must be individually evaluated for eligibility by the Medical Monitor).
* Have a documented pre-Alpha1-Proteinase Inhibitor (PI) augmentation therapy serum alpha-1 antitrypsin (AAT) level <11 micrometer (μM) (80 milligrams per decilitre (mg/dL) if measured by radial immunodiffusion or 50 mg/dL if measured by nephelometry).
* Subjects may be naïve to Alpha1-PI augmentation therapy or may be currently receiving Alpha1-PI augmentation therapy or received Alpha1-PI augmentation therapy within the past. If the subject is currently receiving Alpha1-PI augmentation therapy of any kind, he/she must be willing to discontinue that treatment for at least 25 days prior to the Week 1 (Baseline) Visit and remain off any kind of Alpha1-PI treatment, other than the IPs for this study, while participating in the study.
* At the Screening Visit, have a post-bronchodilator forced expiratory volume (FEV1) ≥30% and <80% of predicted and FEV1/forced vital capacity (FVC) <70% (Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage II or III).

Exclusion Criteria:

* Have had a moderate or severe Chronic obstructive pulmonary disease (COPD) exacerbation during the 4 weeks before the Week 1 (Baseline) Visit.
* Have history of lung or liver transplant.
* Have any lung surgery during the past 2 years (excluding lung biopsy).
* Have severe concomitant disease (example, congestive heart failure, clinically significant pulmonary fibrosis, malignant disease [except for skin cancers other than melanoma], history of acute hypersensitivity pneumonitis reaction, or current chronic hypersensitivity pneumonitis).
* Females who are pregnant, breastfeeding or, if of child-bearing potential, unwilling to practice a highly effective method of contraception (oral, injectable, or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study.
* Have smoked during the past 6 months or a positive urine cotinine test at the Screening Visit that is due to smoking.
* Participate in another Investigational product (IP) study within one month prior to the Week 1 (Baseline) Visit.
* Have history of anaphylaxis or severe systemic response to any plasma-derived Alpha1-PI preparation or other blood product(s).
* Use systemic steroids above a stable dose equivalent to 5 mg/day prednisone (i.e., 10 mg every 2 days) within the 4 weeks prior to the Week 1 (Baseline) Visit. It is recommended to maintain the same dose throughout the study.
* Use systemic or aerosolized antibiotics for a chronic COPD exacerbation within the 4 weeks prior to the Week 1 (Baseline) Visit.
* Have known selective or severe Immunoglobulin A (IgA) deficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 668 days
Number of Participants With Suspected Adverse Drug Reactions (ADRs) | Up to 668 days
Number of Participants With Infusion Site Reactions | Up to 668 days
Number of Participants With Serious Adverse Events (SAEs) | Up to 668 days
Number of Participants With AEs and SAEs Leading to Discontinuation | Up to 668 days
Number of Participants With Chronic Obstructive Pulmonary Disease (COPD) Exacerbations | Up to 668 days
Number of Participants With Clinically Significant Abnormalities in Vital Signs (Heart Rate, Blood Pressure, Respiratory Rate, and Temperature) | Up to 668 days
Change from Baseline in Forced Expiratory Volume in 1 Second (FEV1) | Up to 668 days
Change from Baseline in Forced Vital Capacity (FVC) | Up to 668 days
Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters (Chemistry, Hematology, Urinalysis) | Up to 668 days
Immunogenicity: Number of Participants With Alpha1-PI Antibodies | Treatment Period 1- Single-Dose Week 1; Treatment Period 2- Repeat-Dose Weeks 1 and 9

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina - Children's Hospital, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No